CLINICAL TRIAL: NCT06984848
Title: Effect of Enzymatic-Containing Mouth Spray (Oral7®) on Xerostomia Symptoms, Salivary Flow Rate, and Oral Health-Related Quality of Life in Older Patients: A Randomised Placebo-Control Trial
Brief Title: Effect of Enzymatic-Containing Mouth Spray (Oral7®) on Xerostomia Symptoms, Salivary Flow Rate, and Oral Health-Related Quality of Life in Older Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZAINAB MAT YUDIN (Industry)
Responsible Party: Sponsor-Investigator, ZAINAB MAT YUDIN, Doctor, MBD MARKETING SDN. BHD.
Organization: MBD MARKETING SDN. BHD. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBDMARKETING
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Xerostomia; Geriatric
Keywords: Xerostomia; dry mouth; geriatric; older patient
MeSH Terms: conditions — Xerostomia | interventions — Lactoperoxidase; Glucose Oxidase; Lactoferrin; Muramidase; Calcium; Xylitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Oral7® mouth spray (Experimental): Oral7® mouth spray contains Natural Enzymes (Lactoperoxidase, Glucose Oxidase, Lactoferrin, Lysozyme), Calcium, Xylitol, Aloe Vera, Natural peppermint.
  Interventions: Combination Product: Oral7® mouth spray contains Natural Enzymes (Lactoperoxidase, Glucose Oxidase, Lactoferrin, Lysozyme), Calcium, Xylitol, Aloe Vera, Natural peppermint.
- Control group (No Intervention): The formulation of the placebo mouth spray is derived from distilled water which will be packaging into an identical spray bottle.

INTERVENTIONS:
Combination Product: Oral7® mouth spray contains Natural Enzymes (Lactoperoxidase, Glucose Oxidase, Lactoferrin, Lysozyme), Calcium, Xylitol, Aloe Vera, Natural peppermint. — This study aims to evaluate the effectiveness of an enzymatic-containing mouth spray (Oral7®) on xerostomia symptoms, unstimulated salivary flow rate, and oral health-related quality of life (OHRQoL) in older patients with xerostomia
  Other Names: Oral7®
  Arms: Intervention group: Oral7® mouth spray

SUMMARY:
Background: Xerostomia, or dry mouth, is a prevalent condition among older adults and has significant implications for oral and systemic health. It is associated with impaired chewing, swallowing, and speech, and increases the risk of oral infections, dental caries, and gum disease. Xerostomia may also contribute to malnutrition and aspiration pneumonia.

Objective: This study aims to evaluate the effectiveness of an enzymatic-containing mouth spray (Oral7®) on xerostomia symptoms, unstimulated salivary flow rate, and oral health-related quality of life (OHRQoL) in older patients with xerostomia.

Methods: A single-center, randomized, double-blind, placebo-controlled trial will be conducted at Hospital Universiti Sains Malaysia from August 2025 to July 2026. Eligible participants aged 60 and above with self-reported xerostomia will be randomly assigned to receive either Oral7® Mouth Spray or a placebo spray for four weeks. The primary outcome is the mean change in Summated Xerostomia Inventory (SXI) scores between groups from baseline to post-intervention. Secondary outcomes include changes in unstimulated salivary flow rate using the sialometry technique and OHRQoL measured by the Geriatric Oral Health Assessment Index (GOHAI) at baseline and three months post-intervention. Data will be analyzed using SPSS version 29.

Conclusion: This trial will provide evidence on the efficacy of Oral7® Mouth Spray in alleviating xerostomia symptoms and improving salivary function and oral health-related quality of life in older adults, potentially guiding future clinical management of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above
* Patients with often or always having dry mouth/xerostomia by asking single-item xerostomia question: "How often does your mouth feel dry?" (Adakah mulut anda sering merasakan kekeringan?). The response options were "Never (Tidak Pernah)," "Sometimes (Kadang-kadang)," "Often (Kerap)," or "Always (Sentiasa/Sepanjang masa)."
* Patients who are taking nutrition orally
* Patients who are able to speak
* Patients who are physically fit to take oral spray on their own.

Exclusion Criteria:

* • Patients on salivary substitutes for the past one week

  * Oral condition that required immediate attention such as mucosal or gingival bleeding, orofacial swelling, oral pain and oral ulcer.
  * Patients who are deaf and mute
  * Those with mental disabilities or documented cognitive deficits that would impair their ability to answer questions independently.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1. To compare the mean change in the Summated Xerostomia Inventory (SXI) between older patients with xerostomia taking Oral7® Mouth Spray versus older patients with xerostomia taking placebo mouth spray at baseline and after an intervention duration of 4 | 1 month
  The minimum score for SXI is 5 and the highest score is 15 . The total score of will be calculated into a single continuous scale score which represents the severity of xerostomia; higher scores represent more severe symptoms.

SECONDARY OUTCOMES:
unstimulated whole salivary flow rate | 1 month
  2. To compare unstimulated whole salivary flow rate measurements using sialometry technique between older patients with xerostomia taking Oral7® Mouth Spray versus older patients with xerostomia taking placebo mouth spray at baseline and after an intervention duration of 4 weeks.

OTHER OUTCOMES:
3. To compare changes and differences in the oral health related quality of life (GOHAI) between older patients with xerostomia taking Oral7® Mouth Spray versus older patients with xerostomia taking placebo mouth spray following post study 3 months. | 3 month
  The overall score was calculated by summing up the score of 12 questions and ranged from 0 to 60. The higher the score indicate the more positive oral health quality of life.